CLINICAL TRIAL: NCT03486041
Title: Randomized Controlled Trial of the Comprehensive Behavioral (ComB) Model of Treatment for Trichotillomania
Brief Title: Comprehensive Behavioral (ComB) Model of Treatment for Trichotillomania
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American University (Other)
Collaborators: University of Chicago (Other)
Responsible Party: Principal Investigator, David A. F. Haaga, Professor of Psychology, American University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ComB controlled trial
Record Dates: First submitted 2018-03-15; First posted 2018-04-03 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Trichotillomania
MeSH Terms: conditions — Trichotillomania | interventions — Neuropsychological Tests

STUDY DESIGN:
Intervention Model Description: Immediate ComB and MAC participants will each be assessed at baseline (week 0). ComB will begin weekly therapy sessions, and MAC will receive weekly phone check-ins. All will be assessed at week 6 [mid-treatment] and week 12 [end of controlled phase]. After week 12, ComB enters maintenance and MAC participants start to receive delayed ComB. There is another assessment at week 25 (3-month followup for immediate ComB, post-ComB for MAC) and a final assessment at week 38 (6-month followup for immediate ComB, 3-month followup for MAC).
Who Masked: Outcomes Assessor
Masking Description: The project coordinator at each site will conduct baseline assessments. All later assessments will be conducted by different research assistants, masked to experimental condition of the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- immediate ComB (Experimental): 12 weekly sessions of ComB treatment in individual therapy, following a detailed manual.
  Interventions: Behavioral: Comprehensive Behavior Modification
- Minimal Attention Control (Placebo Comparator): Weekly brief phone call from therapist to check on participant safety, medication changes if any, and recent stressors. After week 12, participants in this arm received delayed ComB [as in the Experimental condition -- 12 weekly sessions of individual therapy for TTM based on ComB model].
  Interventions: Behavioral: Attention

INTERVENTIONS:
Behavioral: Comprehensive Behavior Modification — Behavior therapy approach to BFRBs involving targeted intervention tactics chosen in accordance with the modality of functioning (ex: Sensory, Cognitive.....) seeming to cause the most frequent and problematic urges to engage in the BFRB. Therapist and client work together, using careful assessments including detailed self-monitoring, to determine what behavioral methods will suffice for lasting change.
  Arms: immediate ComB
Behavioral: Attention — Weekly brief calls from therapist to check on safety and clinical status. No focus on TTM.
  Arms: Minimal Attention Control

SUMMARY:
This study will be the first randomized controlled trial of Comprehensive Behavior Modification (ComB) as a treatment of trichotillomania (TTM). ComB treatment (12 weekly sessions, following a manual developed in an earlier treatment development project) will be compared to Minimal Attention Control among adults (N = 42) with TTM.

DETAILED DESCRIPTION:
Treatment based on the ComB model has been influential in the field of body-focused repetitive behaviors (BFRB's), but there is limited empirical research on its efficacy. Our first project (Falkenstein et al., 2016) developed a 12-session manual for ComB and a method for evaluating therapist adherence to the model that can be used reliably and provided encouraging (uncontrolled) data on the effects of ComB through 3-month follow-up.

The proposed project extends the earlier work in two main ways: (a) using random assignment to ComB vs. comparison condition to test whether ComB works better than the passage of time + demand characteristics of being in a TTM study alone; and (b) gathering initial evidence on how ComB works.

Treatment will be conducted at two sites -- Washington, DC (American University and the Behavior Therapy Center of Greater Washington) and Chicago (University of Chicago). Participants in the Minimal Attention Control condition will receive ComB therapy after the post-treatment [week 12] assessment is conducted. Uncontrolled follow-up data will be collected through 3 (MAC condition) or 6 (immediate ComB condition) months after the end of ComB treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older

  * diagnosed with Trichotillomania
  * medication type and dosage [if any] stable for at least 3 months

Exclusion Criteria:

* active suicidality

  --probable bipolar disorder
* probable psychosis

  * other pressing clinical problem requiring immediate treatment
  * current psychotherapy and unable/unwilling to discontinue

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Change in Massachusetts General Hospital Hairpulling Scale | baseline (week 0), week 6, week 12, week 25, week 38
  7-item self-report measure of TTM symptom severity. Score range = 0 to 28. Higher scores = more severe hairpulling symptoms in past week.
Change in National Institute of Mental Health (NIMH) Trichotillomania Severity and Impairment Scales | baseline (week 0), week 6, week 12, week 25, week 38
  interviewer ratings [to be completed by independent evaluator masked to experimental condition] of TTM symptoms and impairment. Scores on the TSS (symptom severity) range 0 to 25, higher scores reflecting more severe symptoms. Scores on the TIS (impairment) range 0 to 10, higher scores reflecting greater impairment associated with hairpulling
Change in Trichotillomania Diagnostic Interview (modified for DSM-5) | baseline (week 0), week 6, week 12, week 25, week 38
  structured diagnostic interview to determine presence/absence of TTM

SECONDARY OUTCOMES:
Alopecia rating | baseline (week 0), week 6, week 12, week 25, week 38
  Masked rater evaluation of hair loss evident in photo taken of most affected pulling site (1 to 7, higher scores reflecting greater hair loss)
Milwaukee Inventory for Subtypes of Trichotillomania-Adult Version [Revised by Keuthen et al.] | baseline (week 0), week 6, week 12, week 25, week 38
  self-report measure of pulling styles, scores ranging from 0 to 72 on Intention subscale and 0-45 on Emotion subscale [higher scores = better fit for that pulling style)
Client Satisfaction Questionnaire | week 6, week 12, week 25, week 38
  self-report measure of treatment satisfaction. Scores range 0 to 32, higher scores reflecting greater satisfaction with services received.
Stop Signal task | baseline (week 0), week 6, week 12
  computer-implemented neurocognitive test of impulsivity vs. ability to inhibit responses. Measured in milliseconds. One indicator is Stop Signal Reaction Time, higher scores reflecting poorer inhibitory control.

CONTACTS AND LOCATIONS:
Locations (1):
- American University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Carlson EJ, Malloy EJ, Brauer L, Golomb RG, Grant JE, Mansueto CS, Haaga DAF. Comprehensive Behavioral (ComB) Treatment of Trichotillomania: A Randomized Clinical Trial. Behav Ther. 2021 Nov;52(6):1543-1557. doi: 10.1016/j.beth.2021.05.007. Epub 2021 Jun 3. PMID 34656205